CLINICAL TRIAL: NCT03242564
Title: A Retrospective Analysis of the Effects of Red Light LED Therapy on Body Contouring
Brief Title: Effects of Red Light LED Therapy on Body Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vevazz, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vev-2017-1
Record Dates: First submitted 2017-07-26; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active Device (Experimental): Active Device: Vevazz LED red light therapy system
  Vevazz LED red light therapy system is a treatment regimen using the Vevazz LED device for fat removal using LED red light therapy.
  Interventions: Device: Vevazz LED

INTERVENTIONS:
Device: Vevazz LED — Vevazz LED red light therapy is a non-invasive dermatological aesthetic treatment for the reduction of circumference of hips, waist and thighs.

SUMMARY:
The purpose of this study is to determine whether red light therapy using LED 650nm red light for body contouring of the waist, hips and thighs is as effective as red light therapy using Laser 635nm red light.

DETAILED DESCRIPTION:
Red light laser therapy using 635nm red light laser technology has previously been shown to cause lipolysis in subcutaneous fat as a non-surgical method to promote weight loss and body contouring. This study hypothesizes that red LED light therapy using 650nm red light LED (light emitting diode) technology produces similar results to the laser device (red LASER 635nm) when preformed using a specified treatment protocol.

Furthermore, it is hypothesized that the Vevazz therapy program achieves the results after a single 28 minute treatment. The predicate 635nm LED device (Photonica Professional by Ward Photonics) achieves its results after one 32 minute therapy program.

The Vevazz therapy program uses the Vevazz LED device for fat removal using LED red light therapy. This multi-site study reviews results from 66 randomly selected patients after a single treatment using the Vevazz LED device.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older.
* May be male or female.
* Generally good health.

Exclusion Criteria:

* Minors.
* Open wounds or sores.
* Pacemaker.
* Photosensitivity.
* Epilepsy.
* Any form of cancer.
* Severe kidney or liver problems.
* Thyroid problems.
* Pregnant or nursing.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Fat Amount (Reduction) in Treatment Area as Measured in Inches Lost | One 28 minute treatment session.
  Circumferential measurement of thighs, hips and waist before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Fettig, Study Director — Owner
Locations (1):
- Vevazz, LLC, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.